CLINICAL TRIAL: NCT03100292
Title: Efficacy and Safety of Bariatric Surgery for Korean Morbidly Obese Patients : Prospective Multicenter Cohort Study
Brief Title: Korean OBEsity Surgical Treatment Study
Acronym: KOBESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Do Joong Park, Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-1608/357-005
Record Dates: First submitted 2017-02-23; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Bariatric Surgery Candidate; Obesity, Morbid
Keywords: primary bariatric surgery; morbid obesity; South Korea; sleeve gastrectomy; Roux-en Y gastric bypass
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bariatric surgery (Experimental): This trial is a single-arm study and the enrolled patients are going to undergo sleeve gastrectomy (SG) or Roux-en-Y gastric bypass (RYGB).
  If the patient has Barrett's esophagus on the preoperative endoscopy, SG is not permitted. Inflammatory bowel disease and Helicobacter pylori infection on a rapid urease test are contraindications of RYGB.
  Interventions: Other: Sleeve gastrectomy or Roux-en-Y gastric bypass

INTERVENTIONS:
Other: Sleeve gastrectomy or Roux-en-Y gastric bypass

SUMMARY:
This trial is a multi-center, single-arm, prospective, observational cohort study of patients undergoing primary bariatric surgical procedures in Korea. A total of 100 patients will be recruited over a 1-year period from 2016 to 2017, and will be followed for a mean follow-up period of 1 year after surgery. The eligible subjects who have given their consent to participate will undergo one of two surgical procedures; sleeve gastrectomy and Roux-en Y gastric bypass.

The primary objective of this clinical trial is to measure the changes in body weight (kg) and waist circumference (cm) of the enrolled patients at postoperative 1 year. Secondary outcomes are improvement or remission rates of obesity-related co-morbidity (hypertension, type 2 diabetes, dyslipidemia, and sleep apnea), and the change in quality of life. Additionally, postoperative incidences of morbidity and mortality, micronutrient status, body composition, and cost-effectiveness of surgical intervention will be examined.

ELIGIBILITY:
Inclusion Criteria:

1. body mass index (BMI) ≥ 35 kg/m2 or BMI ≥ 30 kg/m2 with co-morbidities such as hypertension, glucose intolerance, dyslipidemia, and sleep apnea
2. being suitable for general anesthesia
3. being able to give informed consent and committed to follow-up
4. Female patients should have a negative urine pregnancy test at screening and agree to use reliable method of contraception for 1 year.

Exclusion Criteria:

1. prior bariatric surgery of any kind
2. being unable to understand the risks, benefits and compliance requirements of this trial
3. pregnancy or planning on being pregnancy
4. non-Korean speaker
5. American society of anesthesiology (ASA) class IV or higher
6. malignancy within 5 years.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
body weight (cm) change | postoperative 1-year
waist circumference (cm) change | postoperative 1-year

SECONDARY OUTCOMES:
remission rates of obesity-related co-morbidity (hypertension, type 2 diabetes, dyslipidemia, and sleep apnea) | postoperative 1-year
Quality of life change | postoperative 1-year
  EuroQol-5D (EQ-5D), the impact of weight on QoL (IWQOL) and the obesity-related psychosocial problem scale (OP-scale) are used to assess the improvement of QoL
Morbidity | postoperative 1-year
Mortality | postoperative 1-month
Micronutrients' deficiency | postoperative 1-year
  iron, ferritin, calcium, phosphate, albumin, vit.B12, vit.D, and parathyroid hormone
body composition change | postoperative 1-year
  bioelectrical impedance analysis and fat measurement CT
cost-effectiveness | postoperative 1-year
  cost-utility analysis using lifetime expected costs and quality-adjusted life years (QALYs)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee G, Park YS, Cho C, Lee H, Park J, Park DJ, Lee JH, Lee HJ, Ha TK, Kim YJ, Ryu SW, Han SM, Yoo MW, Park S, Han SU, Heo Y, Jung BH. Short-term changes in the serum metabolome after laparoscopic sleeve gastrectomy and Roux-en-Y gastric bypass. Metabolomics. 2021 Aug 5;17(8):71. doi: 10.1007/s11306-021-01826-y. PMID 34355282
- [Derived] Park YS, Park DJ, Lee JH, Lee HJ, Ha TK, Kim YJ, Ryu SW, Han SM, Yoo MW, Park S, Han SU, Heo Y. Korean OBEsity Surgical Treatment Study (KOBESS): protocol of a prospective multicentre cohort study on obese patients undergoing laparoscopic sleeve gastrectomy and Roux-en-Y gastric bypass. BMJ Open. 2017 Oct 16;7(10):e018044. doi: 10.1136/bmjopen-2017-018044. PMID 29042391